CLINICAL TRIAL: NCT03277651
Title: Developing a Hemodynamics Based Noninvasive Diagnostic Platform for Liver Fibrosis/Cirrhosis and Portal Hypertension
Brief Title: Noninvasive Diagnostic Platform for Liver Fibrosis and Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Hemodynamics Models for CLD
Record Dates: First submitted 2017-09-04; First posted 2017-09-11 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Liver Fibrosis; Cirrhosis; Portal Hypertension
Keywords: noninvasive; Hemodynamics
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver fibrosis: liver biopsy proved
  Interventions: Diagnostic Test: hemodynamics tests
- portal hypertension: hepatic venous pressure gradient (HVPG) proved
  Interventions: Diagnostic Test: hemodynamics tests

INTERVENTIONS:
Diagnostic Test: hemodynamics tests — Hemodynamics tests for intrahepatic blood flow by colour doppler ultrasound

SUMMARY:
This study is to establish a noninvasive diagnostic platform based on hemodynamic information for the assessment of liver fibrosis, liver cirrhosis and portal hypertension.

DETAILED DESCRIPTION:
As the hemodynamics of liver vessels depend on the liver tissue mechanics, we hypothesize that the hemodynamics measurements of the liver are strongly correlated with the stages of liver fibrosis and portal hypertension, and can therefore serve as an alternative means of diagnosis. We have developed a physics-based mathematical model that incorporates our biological understanding of fibrosis development. The model quantitatively predicts changes of liver tissue stiffness and blood flow dynamics as a function of fibrosis stage. Preliminary data using ultrasound Doppler images and needle biopsy from liver fibrosis patients have suggested the 'prove of principle. We propose further test our hypothesis by collecting and analyzing ultrasound Doppler and biopsy data to confirm the correlation between blood flow dynamics and disease stage from patients with hepatic fibrosis and portal hypertension. If tested true, we can expect to use features of ultrasound Doppler as a non-invasive means of diagnosis for fibrosis and portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who undergo liver biopsy or hepatic venous pressure gradient test

Exclusion Criteria:

* decompensated liver diseases (including ascites, variceal bleeding or hepatic encephalopathy);
* alpha-fetoprotein >100 ng/ml or serum creatinine >1.5 × upper limit of normal (ULN);
* any malignant tumor;
* any complications of severe heart, lung, kidney, brain, blood diseases or other important systematic diseases;
* severe neurological or psychological disease;
* pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients who undergo liver biopsy or hepatic venous pressure gradient test in Zhongshan hospital Fudan University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | baseline
  Diagnostic power of the hemodynamics based noninvasive platform for liver fibrosis or portal hypertension
Specificity | baseline
  Diagnostic power of the hemodynamics based noninvasive platform for liver fibrosis or portal hypertension
Positive predictive value (PPV) | baseline
  Diagnostic power of the hemodynamics based noninvasive platform for liver fibrosis or portal hypertension
Negative predictive value (NPV) | baseline
  Diagnostic power of the hemodynamics based noninvasive platform for liver fibrosis or portal hypertension
Area under ROC curve (AUROC) | baseline
  Diagnostic power of the hemodynamics based noninvasive platform for liver fibrosis or portal hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zheng L, Shi N, Li P, Ge H, Tu C, Qu Y, Wang Y, Lin Y, Chen S, Sun D, Weng C, Wu S, Jiang W. Development and validation of machine learning models to predict esophagogastric variceal rebleeding risk in HBV-related cirrhosis after endoscopic treatment: a prospective multicenter study. EClinicalMedicine. 2025 Aug 20;87:103436. doi: 10.1016/j.eclinm.2025.103436. eCollection 2025 Sep. PMID 40896458